CLINICAL TRIAL: NCT02164825
Title: Comparison Between Single-shot Femoral Nerve Block and Epidural Techniques for Total Knee Arthroplasty: a Randomized Controlled Trial
Brief Title: Total Knee Arthroplasty Analgesia: Single-shot Femoral Nerve Block or Epidural?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Hospitalar do Tâmega e Sousa (Other)
Responsible Party: Principal Investigator, Mariana Marques da Cunha, MD, Centro Hospitalar do Tâmega e Sousa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CHTSA001
Record Dates: First submitted 2014-06-05; First posted 2014-06-17 (Estimated); Last update posted 2015-02-05 (Estimated); Status verified 2014-06

CONDITIONS: Postoperative Pain Treatment for Total Knee Arthroplasty
MeSH Terms: interventions — Morphine; Ropivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Single-shot nerve block (Experimental): Efficacy compared to epidural
  Interventions: Drug: Ropivacaine perineural injection
- Continuous epidural (Active Comparator): Continuous epidural perfusion
  Interventions: Drug: morphine and ropivacaine

INTERVENTIONS:
Drug: Ropivacaine perineural injection — Ultrasound guided single-shot femoral nerve block
  Arms: Single-shot nerve block
Drug: morphine and ropivacaine — Continuous epidural analgesic perfusion Epidural perfusion with morphine and ropivacaine.
  Arms: Continuous epidural

SUMMARY:
Single-shot femoral nerve block is similar to continuous epidural technique for postoperative analgesia in total knee arthroplasty

ELIGIBILITY:
Inclusion Criteria:

* Elective total knee arthroplasty

Exclusion Criteria:

* Coagulopathy
* Neuropathy
* Morbid obesity
* local anesthetics allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-01; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Pain Score on the numeric pain score | 48 hours
  Patients will be evaluated at 48 hours. At these time frame pain score at rest and during movement will be accessed.

SECONDARY OUTCOMES:
Side effects as a measure of safety and tolerability | 48 hours
  Side effects of both interventions. Number of patients with side effects like nausea, vomiting, hypotension and pruritus.
Rescue analgesic consumption. | 48 hours
  Opioid rescue needs in the first 48 hours after surgery.
Patients satisfaction. | 48 hours
  Evaluation of patient´s satisfaction with pain control (asking the patient to classify the grade of satisfaction).

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Hospitalar Tâmega e Sousa, Penafiel, Penafiel, Portugal